CLINICAL TRIAL: NCT02749071
Title: A Multicenter, Randomized, Double-Blind, Sham-Controlled Clinical Investigation of the EndoStim® Lower Esophageal Sphincter (LES) Stimulation System for the Treatment of Gastroesophageal Reflux Disease (GERD)
Brief Title: An Investigation of the EndoStim® Lower Esophageal Sphincter (LES) Stimulation System for the Treatment of Reflux
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company no longer operational
Sponsor: EndoStim Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS-100
Record Dates: First submitted 2016-04-15; First posted 2016-04-22 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Gastroesophageal Reflux Disease (GERD); Reflux, Gastroesophageal; Gastroesophageal Reflux; Acid Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Sham Comparator): This group will undergo laparoscopic implantation surgery. The device will not be activated: Sham EndoStim stimulation for first six months of study. It will be activated at the Month 6 visit and provide lower esophageal stimulation from Month 6 thru end of study.
  Interventions: Procedure: Laparoscopic implantation surgery; Device: EndoStim stimulation from Month 6 thru end of study; Device: Sham EndoStim stimulation for first six months of study
- Treatment Group (Experimental): The group will undergo laparoscopic implantation surgery. The device will be activated two weeks post-implantation and the subject will receive EndoStim stimulation for first six months of study and continue with EndoStim stimulation from Month 6 thru end of study.
  Interventions: Procedure: Laparoscopic implantation surgery; Device: EndoStim stimulation for first six months of study; Device: EndoStim stimulation from Month 6 thru end of study

INTERVENTIONS:
Procedure: Laparoscopic implantation surgery — Laparoscopic surgery to implant the pulse generator and bipolar lead.
Device: EndoStim stimulation for first six months of study — Lower esophageal stimulation
  Other Names: EndoStim Implantable Pulse Generator (IPG); lower esophageal stimulation
  Arms: Treatment Group
Device: EndoStim stimulation from Month 6 thru end of study — Lower esophageal stimulation
  Other Names: EndoStim Implantable Pulse Generator (IPG); lower esophageal stimulation
Device: Sham EndoStim stimulation for first six months of study — EndoStim device remains "off" (no stimulation delivered)
  Arms: Control Group

SUMMARY:
The purpose of this investigation is to demonstrate the safety and effectiveness of Lower Esophageal Sphincter (LES) Stimulation System in treating gastroesophageal reflux disease (GERD). This investigation is a multicenter, randomized, double-blind, sham-controlled study. After the implant procedure, subjects will be randomized to either the Treatment Group (immediate stimulation) or Control Group (delayed stimulation) for six months followed by an additional open-label phase in which all subjects will receive electrical stimulation. Subjects continue on stimulation treatment in an extended open-label follow-up phase through 5 years post-stimulation.

DETAILED DESCRIPTION:
The purpose of this investigation is to demonstrate the safety and effectiveness of the EndoStim® Lower Esophageal Sphincter (LES) Stimulation System in the treatment of subjects with gastroesophageal reflux disease (GERD). This investigation is a multicenter, randomized, double-blind, sham-controlled clinical investigation. After the implant procedure, subjects will be randomized to either the Treatment Group (immediate stimulation) or Control Group (delayed stimulation) for a 6-month, double-blind phase followed by an additional open-label treatment phase in which all subjects will receive electrical stimulation therapy for a total of 12 months. Subjects continue on stimulation treatment and an extended open-label follow-up phase includes an 18 month post-stimulation phone interview followed by annual visits through 5 years post-stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent
2. Able and willing to comply with required study procedures and follow-up schedule
3. 22 - 75 years of age at the time of informed consent
4. Documented symptoms of gastroesophageal reflux disease (GERD) for longer than 6 months (regurgitation and/or heartburn which is defined as burning epigastric or substernal pain which responds to acid neutralization or suppression) which requires daily use of proton pump inhibitors (PPIs) or other anti-reflux drug therapy, who continue to have symptoms despite maximum medical therapy or are "intolerant" -severe side-effects (e.g. anaphylaxis or severe allergic reaction, recurrent C. difficile, severe hypomagnesaemia) to one PPI or mild/moderate side effect (e.g. nausea, vomiting, diarrhea or abdominal pain) to at least 2 PPIs of different chemical classes.
5. Symptomatic improvement on PPI therapy demonstrated by a composite GERD-health-related quality of life (HRQL) score of ≥20 off PPI, and a ≥10 point improvement on PPI compared to the off PPI composite GERD-HRQL score. Patients who meet the definition above of PPI intolerant are not required to have ≥10 point improvement. The on-PPI score to satisfy this criterion will be the score from the GERD-HRQL assessment completed after resuming PPIs following the Baseline visit.
6. Excessive lower esophageal acid exposure during pH monitoring (defined as distal esophageal pH < 4 for > 6.0% of the monitoring time) performed after at least 5 days off of PPIs and at least 2 days off of H2 blockers. At least 18 hour of esophageal pH recording will be considered adequate and inclusion will be based on the day (at least 18 hours of valid data) with the highest acid exposure percentage time.
7. Esophagitis ≤ Grade B (Los Angeles (LA) classification) as measured by upper endoscopy off PPI and H2 blockers for 10-14 days
8. Esophageal body contraction amplitude > 30 mmHg for > 30% of swallows and > 30% peristaltic contractions on HRM or ≥ 30% peristaltic contractions with DCI >450.
9. Suitable surgical candidate able to undergo general anesthesia and laparoscopic surgery

Exclusion Criteria:

1. Previous EndoStim LES System implant and/or implant attempt
2. Previous surgery involving the gastroesophageal junction or the lead implant site, such as a Nissen fundoplication
3. Previous endoscopic intervention for the treatment of GERD and/or Barrett's esophagus
4. Hiatal hernia larger than 3 cm as determined by endoscopy
5. History of gastroparesis
6. Any non-GERD esophageal motility disorders that in the opinion of investigator precludes an anti-reflux procedure
7. History of or known esophageal stricture or significant esophageal anatomic abnormalities (obstructive lesions, etc.)
8. Barrett's esophagus or any grade of dysplasia
9. Documented history of esophagitis Grade C or D (LA Classification)
10. History of suspected or confirmed esophageal or gastric cancer
11. Esophageal or gastric varices
12. Symptoms of dysphagia more than once per week every week within the last 3 months
13. Unable to tolerate withdrawal from H2 Blockers or PPI medications
14. Suspected or known allergies to titanium, platinum, iridium, stainless steel, silicone, epoxy, or nylon
15. Body mass index (BMI) > 35 kg/m2
16. Any significant multisystem diseases
17. Autoimmune or a connective tissue disorder (scleroderma, dermatomyositis, Calcinosis-Raynaud's-Esophagus Sclerodactyly Syndrome (CREST), Sjogren's Syndrome, Sharp's Syndrome, etc.) requiring therapy in the preceding 2 years
18. Type 1 diabetes mellitus or uncontrolled Type 2 diabetes mellitus (T2DM) defined as HbA1c > 9.5 in the previous 6 months or at screening/baseline
19. Significant cardiac arrhythmia or ectopy or significant cardiovascular disease (i.e. unstable angina pectoris, hemodynamically significant valvular disease, severe congestive heart failure), or any cardiac therapeutic intervention within the last 6 months.
20. Significant cerebrovascular event within the last 6 months
21. Existing implanted electrical stimulator (pacemaker, implantable cardioverter defibrillator, deep brain stimulator (DBS), bone growth or pelvic floor stimulators, drug pumps, etc.)
22. Female subject of child-bearing potential and is pregnant or nursing, or intends to become pregnant during the trial period, who is not using a reliable form of birth control
23. Currently enrolled in other potentially confounding research
24. Active infection as determined by the investigator
25. History of any malignancy, other than basal cell carcinoma, in the last 2 years
26. Life expectancy less than 3 years aa. Diagnosed major psychiatric disorder (bipolar, schizophrenia, etc.) bb. Any condition that, at the discretion of the investigator or sponsor, would interfere with accurate interpretation of the study endpoints or preclude participation in the trial

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2016-05; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Rate of device and/or procedure-related serious adverse events | 12 months
  Rate of occurrence of device and/or procedure-related serious adverse events after 12 months
Percentage of subjects achieving pH success (pH<4 for mo more than 5.3% of time or at least 50% improvement in pH compared to baseline) | Comparison of 6 months to baseline data
  Comparison between treatment and control group: percentage of subjects achieving pH success ((pH<4 for mo more than 5.3% of time or at least 50% improvement in pH compared to baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Shaheen, MD, MPH, Principal Investigator — University of North Carolina
Locations (21):
- United States (18):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - HonorHealth Research Institute, Scottsdale, Arizona
  - University of Southern California (USC), Los Angeles, California
  - Stanford Center for Clinical Research, Stanford, California
  - Institute of Esophageal and Reflux Surgery, Englewood, Colorado
  - University of South Florida, Tampa, Florida
  - Cornell University Weill Medical College, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas HealthCare System, Charlotte, North Carolina
  - The MetroHealth System, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Oregon Clinic, Portland, Oregon
  - Oregon Health Science University, Portland, Oregon
  - Allegheny Health Network Research Institute, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Scott & White Research Institute, Round Rock, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium
- Clinical Trial Center Maastricht, Maastricht, Netherlands
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study website — http://www.lessgerd.com